CLINICAL TRIAL: NCT01554969
Title: Phase I Trial of Ganetespib, Capecitabine, and Radiation in Rectal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Synta Pharmaceuticals Corp. (Industry)
Responsible Party: Principal Investigator, Bassel El-Rayes, Principal Investigator, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00054181; STA 9090 (Other: Other)
Record Dates: First submitted 2012-03-13; First posted 2012-03-15 (Estimated); Last update posted 2016-02-22 (Estimated); Status verified 2016-02

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms | interventions — Capecitabine; STA 9090

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- capecitabine + ganetespib . (Experimental): Capecitabine oral medication. Ganetespib IV medication
  Interventions: Drug: capecitabine + ganetespib

INTERVENTIONS:
Drug: capecitabine + ganetespib — Capecitabine will be started on Day 1 of the concurrent chemo-radiation phase at the specified dose, and is given orally twice daily for the entire duration of radiation therapy.
  Ganetespib will be started on Day 1 of radiation therapy and is administered as IV infusion over 1 hour on days 1, 8, 15 for cycle 1 and then on days 29 and 36 for cycle 2.
  In all patients, ganetespib monotherapy will be given up to 2 weeks prior to start of concurrent chemoradiation. Sequential biopsies will be taken at baseline and prior to the start of concurrent chemoradiation. In the dose escalation part of the study, the starting does of ganetespib is 60mg/m² once weekly, and capecitabine at a dose of 825 mg/m² twice daily.
  Other Names: Ganetespib; STA-9090

SUMMARY:
The purpose of this study is to find out what effects, good and/or bad, the combination of the study drug, capecitabine, and radiation have on you and your cancer. Capecitabine, radiation, and the study drug kill cancer cells in different ways. Giving these treatments together may make your cancer shrink or slow down its growth more than it would if you got treated with capecitabine and radiation alone.

This is a Phase I drug study of ganetespib given together with capecitabine and radiation in patients with locally advanced rectal cancer. Ganetespib is an experimental drug; not approved by the Food and Drug Administration (FDA). The other two, capecitabine and radiation, are approved by FDA for use in rectal cancer.

In this study, the investigators will test different dosages of the "investigational" (experimental) drug, called ganetespib (the study drug). The study drug is "investigational" because it is not approved by the FDA for use. The study drug has been previously tested in humans. The study uses a well-established process of slowly increasing drug dosage to determine the highest dosage that can be given without causing serious side effects. In addition, the study will help researchers to determine what the side effects and drug interactions might be.

The study will also look at the drug's pharmacokinetics (PK). PK is how the study drug and capecitabine with radiation work in your body (for example how long the drugs last in your body.)

DETAILED DESCRIPTION:
Patients with rectal cancer who meet the eligibility criteria will be offered to enroll on the study. As part of the study patients will receive the standard of care capecitabine (825 mg/m² by mouth twice daily) and radiation. Patients will start on ganetespib (STA9090) at a set dose level.

The treatment consists of two parts. In the first part patients will receive ganetespib at full dose twice a week through the vein for two weeks. At the end of two weeks, a biopsy of the tumor will be performed to evaluate the effect of the drug on the tumor. In the second phase, patients will receive capecitabine, radiation and ganetespib at a specified dose level for 5 to 6 weeks. After completion of this phase, patients will have surgery to remove the tumor. Each three patients will be treated at a specified dose level. Patients will be monitored at least once a week for side effects. If there are no side effects in three consecutive patients, then the investigators will treat the next three patients at a higher dose level.

ELIGIBILITY:
Inclusion Criteria:

* Must be at least 18 years of age
* Stage II or III histologically-proven rectal adenocarcinoma. The distal border of the tumor must be at or below the peritoneal reflection, defined as within 12 centimeters of the anal verge by proctoscopic examination.
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0 or 1
* Adequate hematologic function as defined by:

  * Absolute neutrophil count ≥ 1,500 cells/µL
  * Platelets ≥ 100,000/µL
  * Hemoglobin ≥ 9.0g/dL
* Adequate hepatic function as defined by:

  * Total bilirubin ≤ 1.5 x the upper limit of normal (ULN)
  * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 x ULN
  * Albumin ≥ 3.0 g/dL
* Adequate renal function as defined by:

  * Serum creatinine ≤ 1.5 x ULN
  * Calculated creatinine clearance of ≥ 50 mL/min
* International normalized ratio (INR) ≤ 1.5. Anticoagulation is allowed only with low molecular weight heparin (LMWH). Patient receiving LMW heparin on stable therapeutic dose for more than 2 weeks or with factor Xa level < 1.1 U/mL are allowed on the trial.
* Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures
* Ability to understand and willingness to sign a written informed consent document
* Female subjects of childbearing potential and males must agree to use adequate contraception (e.g., hormonal or barrier method of birth control; abstinence) for the duration of study treatment
* Female subjects of childbearing age must have a negative serum pregnancy test at study entry.

Exclusion Criteria:

* History of previous radiation therapy to the abdomen or pelvis
* History of previous chemotherapy for rectal cancer
* Major surgery within 4 weeks prior to first dose of ganetespib
* Poor venous access for study drug administration. The study drug must be administered via peripheral venous access or through vascular access devices (VADs) (such as ports and peripherally-inserted central catheters [PICCS] containing silicone catheters. Use of VADs with catheters made of any other material is not allowed.
* History of severe allergic or hypersensitivity reactions to excipients (e.g., Polyethylene glycol [PEG] 300 and Polysorbate 80)
* Baseline corrected QT interval (QTc) > 450 msec or previous history of QT prolongation while taking other medications
* Ventricular ejection fraction (Ef) ≤ 55% at baseline
* Treatment with chronic immunosuppressants (e.g., cyclosporine following transplantation)
* Women who are pregnant or lactating
* Uncontrolled intercurrent illness
* Other medications, or severe acute/chronic medical or psychiatric condition, or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, and in the judgment of the investigator would make the subject inappropriate for entry into this study
* Patients must be able to take oral medications.
* Unequivocal metastatic disease on computed tomography or chest X-ray
* Clinically significant comorbid conditions such as cardiovascular disease or significant peripheral vascular (e.g., uncontrolled hypertension, myocardial infarction, unstable angina) within 6 months of study entry, serious cardiac arrhythmia requiring medication, and uncontrolled infection.
* Clinical evidence of bleeding diathesis or coagulopathy
* Significant involvement of the bladder by the tumor
* Patients with prior malignancies, including pelvic cancer, are eligible if they have been disease free for > 5 years. Patients with prior in situ carcinomas are eligible provided there was complete removal.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2012-05; Primary Completion 2015-03 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Tumor response and disease progression will be evaluated in this study using the international criteria proposed by the Response Evaluation Criteria in Solid Tumors (RECIST). | 8 weeks
  Changes in only the largest diameter (unidimensional measurement) of the tumor lesions are used in the RECIST criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Bassel El-Rayes, MD, Principal Investigator — Emory University
Locations (1):
- Emory University Winship Cancer Institute, Atlanta, Georgia, United States

REFERENCES:
- [Derived] Nagaraju GP, Park W, Wen J, Mahaseth H, Landry J, Farris AB, Willingham F, Sullivan PS, Proia DA, El-Hariry I, Taliaferro-Smith L, Diaz R, El-Rayes BF. Antiangiogenic effects of ganetespib in colorectal cancer mediated through inhibition of HIF-1alpha and STAT-3. Angiogenesis. 2013 Oct;16(4):903-17. doi: 10.1007/s10456-013-9364-7. Epub 2013 Jul 10. PMID 23838996